CLINICAL TRIAL: NCT01276340
Title: Prospective Evaluation of Keat Electrostimulator in the Auto-reeducation
Brief Title: Prospective Evaluation of Keat Electrostimulator in the Auto-reeducation of Female Urinary Incontinence
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 1008433
Record Dates: First submitted 2011-01-11; First posted 2011-01-13 (Estimated); Last update posted 2012-05-17 (Estimated); Status verified 2012-05

CONDITIONS: Urinary Incontinence
Keywords: Urinary Incontinence; Urinary stress incontinence; Urinary urge incontinence; Women; electrical stimulation; KEAT stimulator; quality of life
MeSH Terms: conditions — Urinary Incontinence; Urinary Incontinence, Stress; Urinary Incontinence, Urge

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: women with urinary incontinence
  Interventions: Device: KEAT stimulator

INTERVENTIONS:
Device: KEAT stimulator — electrical stimulation with KEAT stimulator : 4 times per week during 2 months

SUMMARY:
The investigators performed a prospective analysis of 450 women with stress, urge and mixed incontinence in order to assess the health-related quality of life (Contilife® questionnaire) and the objective cure rate after two months of electrical stimulation (Keat® stimulator). Management of urinary incontinence with the Keat® stimulator could given an improvement in the quality of life and a good rate of satisfaction without side effect.

Objective cure is as good as subjective improvement especially in urinary stress incontinence. Keat® stimulator is a non-invasive and simple new technique that could be the bew first-line non surgical treatment for female urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

* women
* age > 18 years
* stress, urge or mixed incontinence with indication of perineal reeducation
* follow in gynecology

Exclusion Criteria:

* incontinence due to neurological disorders
* younger than 18 years old
* pregnancy
* patient with pace-maker
* patient with gynecological cancer
* patient who don't understand the electrical stimulation procedure

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women with stress, urge and mixed incontinence with an indication for perineal reeducation follow in gynecology
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2010-09; Primary Completion 2011-12 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
change of quality of life after electrostimulation | 2 months
  Change from baseline in quality of life after 2 months of electrostimulation Measurement of health-related quality of life with "contilife" questionnaire

SECONDARY OUTCOMES:
change of urinary handicap after electrostimulation | 2 months
  Change from baseline in urinary handicap after 2 months of electr-st-imulation. Measurement of urinary handicap with "MHU" questionnaire
satisfaction after electrostimulation | 2 months
  description of patient's satifaction 2 months after electrostimulation by satisfaction questionaire

CONTACTS AND LOCATIONS:
Overall Officials: Gautier CHENE, MD, Principal Investigator — CHU de Saint-Etienne
Locations (6):
- France (6):
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - CHU Dijon, Dijon
  - CHU Grenoble, Grenoble
  - CH Issoire, Issoire
  - CHU Limoges, Limoges
  - Hospices Civils de Lyon, Lyon